CLINICAL TRIAL: NCT01203956
Title: A Multi Center, Prospective, Randomized, Double Blind, Crossover Study to Compare the DeVilbiss AutoAdjust With and Without the Smartflex Device Modification; "AutoAdjust With SmartFlex Study"
Brief Title: DeVilbiss AutoAdjust With SmartFlex Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeVilbiss Healthcare LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DHC-C001
Record Dates: First submitted 2010-08-31; First posted 2010-09-17 (Estimated); Results first posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: AutoAdjust; SmartFlex; Apnea Hypopnea Index; Patient reported outcomes
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Reference Standards

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SmartFlex (Experimental): Use Continuous Airway Pressure device with SmartFlex engaged
  Interventions: Device: SmartFlex
- Standard (Active Comparator): Use Continuous Airway Pressure device without SmartFlex engaged
  Interventions: Device: Standard

INTERVENTIONS:
Device: SmartFlex — Device used with smartflex engaged.
  Other Names: DeVilbiss AutoAdjust with SmartFlex
  Arms: SmartFlex
Device: Standard
  Other Names: DeVilbiss AutoAdjust without SmartFlex
  Arms: Standard

SUMMARY:
There will be equivalent therapeutic effectiveness between SmartFlex and standard modes when using the DeVilbiss AutoAdjust device.

ELIGIBILITY:
Inclusion Criteria:

* Epworth Sleepiness Scale >10
* Body Mass Index > 26
* Apnea-hypopnea index (AHI) ≥15 (mod to severe range)
* AHI ≤ 10 at therapeutic continuous positive airway pressure (CPAP) pressure
* CPAP naïve patients
* Polysomnogram (PSG) within 3 months of enrollment
* Average oxygen saturation by pulse oximetry (SpO2) > 90% during titration
* Sleep efficiency on titration night ≥ 78%

Exclusion Criteria:

* Diagnosis of mild obstructive sleep apnea (OSA)
* Co-morbid conditions which render participation to be at risk these may include patients with congestive heart failure, chronic obstructive pulmonary disease (COPD) or psychiatric illness
* Allergies to mask materials
* Difficulties with nasal breathing
* Evidence of another primary sleep disorder
* Evidence of arousing periodic limb movements during titration
* Contraindications as listed on product labeling.
* Pregnant
* Currently diagnosed with depression if symptomatic
* Predominately central sleep apnea
* Deemed medically unsuitable by investigator
* Evidence of any type of infection or treatment of an infectious condition during the period of research participation
* Full Face Mask during titration
* Have a bi-level requirement
* CPAP pressure >15cmH2O
* Subjects with tracheotomy
* Uncontrolled hypertension
* Require supplemental oxygen
* Stimulants, major tranquillizers or antipsychotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Rosenthal, MD, Principal Investigator — Sleep Medicine Associates of Texas
Locations (2):
- United States (2):
  - Sleep Medicine Associates of Texas, Dallas, Texas
  - Sleep Therapy and Research Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- SmartFlex First, Then Standard: First two weeks with Smartflex engaged, second two weeks without Smartflex engaged
- Standard First, Then Smartflex: First two weeks without Smartflex engaged, second two weeks with Smartflex engaged
Period: First Two-week Period
Arm/Group | SmartFlex First, Then Standard | Standard First, Then Smartflex
Started | 15 | 13
Completed | 15 (All participants continued to the second two-week period, whether or not they had evaluable results.) | 13 (All participants continued to the second two-week period, whether or not they had evaluable results.)
Not Completed | 0 | 0
Period: Second Two-week Period
Arm/Group | SmartFlex First, Then Standard | Standard First, Then Smartflex
Started | 15 | 13
Attended Sleep Studies for 14 Nights | 15 | 13
Completed | 10 (Completed with evaluable results, as assessed over both two-week study periods.) | 7 (Completed with evaluable results, as assessed over both two-week study periods.)
Not Completed | 5 | 6
Not completed — Non-compliant: no evaluable results | 5 | 6

BASELINE CHARACTERISTICS:
Population: Compliant participants completing study with evaluable results
Groups:
- All Evaluable Subjects: All subjects completing both two-week periods of crossover study, with evaluable results for each period.
Arm/Group | All Evaluable Subjects
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
AHI (apnea-hypopnea index) [Mean (Standard Deviation); unit: events / hour] | 39.8 (21.5)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index (AHI)
Description: Number of apnea/hypopnea events per hour, measured by SmartLink component of device.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: events / hour
Groups:
- SmartFlex: Used CPAP device with SmartFlex engaged, in either first or second two-week period.
- Standard: Used CPAP device without SmartFlex engaged, in either first or second two-week period.
Arm/Group | SmartFlex | Standard
Number analyzed (Participants) | 17 | 17
events / hour | 5.92 (3.75) | 5.56 (3.27)

2. Secondary Outcome: Key Measures That Will be Used to Evaluate the Intervention(s)
Description: The Epworth Sleepiness Scale will be used to evaluate sleepiness The Sleep Wake Activity Inventory will be used to evaluate sleepiness Daily diaries will be used to evaluate daily use of the device
Time Frame: 2 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- SmartFlex: CPAP device used with SmartFlex engaged, either in first or second two-week period.
- Standard: CPAP device used without SmartFlex engaged, either in first or second two-week period.
- EG002: From data available it cannot be determined which mode the subject was using at the time of this event.
Arm/Group | SmartFlex | Standard | EG002
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 4/17 | 4/17 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmartFlex (N=17) | Standard (N=17) | EG002 (N=17)
Uncomfortable breathing due to expiratory resistance (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Mouth breathing which may worsen snoring or OSA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Nasal, sinus or middle ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 1 (1)
Redness on bridge of nose (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatal hernia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Jaw pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pressure sore on bridge of nose (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No